CLINICAL TRIAL: NCT06092801
Title: Development and Validation of Artificial Intelligence Prediction Models Based on Multimodal, Non-contact Captured Information in Predicting Coronary Artery Disease
Brief Title: Prediction of Coronary Artery Disease Based on Multimodal, Non-contact Information With Artificial Intelligence
Status: Completed | Type: Observational
Sponsor: China National Center for Cardiovascular Diseases (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2022-GSP-QN-10
Record Dates: First submitted 2023-10-16; First posted 2023-10-23 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Individuals suspected of coronary artery disease: Individuals suspected of coronary artery disease and referred for evaluation
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
The goal of this observational study are 1) to assess the effectiveness of modalities and/or their combination of multimodal non-contact information in predicting coronary artery disease; 2) to prospectively validate the performance of the developed artificial Intelligence models in predicting coronary artery disease.

DETAILED DESCRIPTION:
This observational study aims to assess the effectiveness and potential mechanism of modalities of non-contact captured bio-physiological information, including facial RGB information, infrared thermography temperature information, gait information, and wearable device information, individually and/or in combination, in predicting coronary artery disease (CAD) with artificial intelligence technology.

Individuals suspected of CAD and referred for evaluation will be invited to participate in the current study for analyzing the non-contact information and association with underlying CAD status, in order to establish the most efficient artificial Intelligence modeling strategy, and prospectively validate the predictive performance of the developed artificial Intelligence models for CAD prediction.

ELIGIBILITY:
Inclusion Criteria:

* Suspected individuals referred to for coronary angiography or coronary computer tomography angiography.

Exclusion Criteria:

* Prior percutaneous coronary intervention (PCI)
* Prior coronary artery bypass graft (CABG)
* Undergoing confirmatory coronary evaluation as pre-operation routines for other cardiac diseases
* With artificial body alteration (e.g. cosmetic surgery, facial trauma, or make-up) that may affect the non-contact information of study interest
* Age less than 18 years old
* Other circumstances that prevent participants from cooperating with the study process
* Decline to consent for study participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Individuals suspected of coronary artery disease and referred for confirmatory evaluation
Sampling Method: Non-Probability Sample
Enrollment: 2978 (Actual)
Dates: Start 2023-11-20 (Actual); Primary Completion 2025-04-09 (Actual); Study Completion 2025-04-09 (Actual)

PRIMARY OUTCOMES:
Sensitivity of algorithm | At the end of enrollment (1 mouth)
  Sensitivity of algorithm in predicting coronary artery disease assessed in test group
Specificity of algorithm | At the end of enrollment (1 mouth)
  Sensitivity of algorithm in predicting coronary artery disease assessed in test group

SECONDARY OUTCOMES:
Area under receiver operating curve (AUC) | At the end of enrollment (1 mouth)
  Area under receiver operating curve of algorithm in predicting coronary artery disease assessed in test group

OTHER OUTCOMES:
Positive predictive value (PPV) of algorithm | At the end of enrollment (1 mouth)
  Positive predictive value (PPV) of algorithm in predicting coronary artery disease assessed in test group
Negative predictive value (NPV) | At the end of enrollment (1 mouth)
  Negative predictive value (NPV) of algorithm in predicting coronary artery disease assessed in test group
Diagnostic accuracy rate | At the end of enrollment (1 mouth)
  Diagnostic accuracy rate of algorithm in predicting coronary artery disease assessed in test group

CONTACTS AND LOCATIONS:
Overall Officials: Shen Lin, M.D., Ph.D., Principal Investigator — Chinese Academy of Medical Sciences, Fuwai Hospital
Locations (1):
- Fuwai Hospital, Chinese Academy of Medical Sciences and Peking Union Medical College, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lin S, Li Z, Fu B, Chen S, Li X, Wang Y, Wang X, Lv B, Xu B, Song X, Zhang YJ, Cheng X, Huang W, Pu J, Zhang Q, Xia Y, Du B, Ji X, Zheng Z. Feasibility of using deep learning to detect coronary artery disease based on facial photo. Eur Heart J. 2020 Dec 7;41(46):4400-4411. doi: 10.1093/eurheartj/ehaa640. PMID 32818267